CLINICAL TRIAL: NCT00566384
Title: Multi-center, Double-blind, Placebo-controlled Study to Investigate the Efficacy and Safety of Daily Oral 100 mg Dehydroepiandrosterone (DHEA) Over 6 Treatment Cycles as a Concomitant Therapy to Oral Contraceptives (OC) to Alleviate Complaints of Reduced Libido in Women With Acquired Female Sexual Dysfunction (FSD) Associated With OC-use
Brief Title: Efficacy and Safety of Oral Dehydroepiandrosterone as a Concomitant Therapy to Oral Contraceptives in Women Complaining of Reduced Libido
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 91692; 310741 (Other: Company Internal); 2006-004397-27 (EudraCT Number)
Record Dates: First submitted 2007-11-29; First posted 2007-12-03 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Libido
Keywords: Loss of libido; Acquired, oral contraceptive -associated female sexual dysfunction
MeSH Terms: interventions — Dehydroepiandrosterone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Active Comparator)
  Interventions: Drug: Dehydroepiandrosterone, BAY86-5314
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dehydroepiandrosterone, BAY86-5314 — Treatment with daily oral intake of two capsules containing 50 mg DHEA each. Treatment duration will be 24 weeks
  Arms: Arm 1
Drug: Placebo — Treatment with daily oral intake of two capsules containing Placebo. Treatment duration will be 24 weeks
  Arms: Arm 2

SUMMARY:
The purpose of the study is to evaluate the effectiveness of the study drug on the libido (sexual desire) of women who are taking oral contraceptives and who have experienced libido reductions as a side-effect of this contraceptive method The hypothesis is that there is superiority in the change in sexual desire and arousal component scores of the FSFI questionnaire from baseline to cycle 6 of the treatment with the study drug as compared to Placebo.

ELIGIBILITY:
Inclusion Criteria:

* Treatment with a oral contraceptive (OC) for at least 3 months and willing to continue the OC
* Loss of libido
* Sexual relationship with a sexually competent partner

Exclusion Criteria:

* Female sexual dysfunction other than HSDD, arousal and orgasmic disorder, such as sexual aversion/phobic disorder, sexual pain disorder/dyspareunia
* Hyperandrogenemic conditions, such as congenital adrenal hyperplasia (CAH), polycystic ovary syndrome (PCOS), Cushing's syndrome or signs of hyperandrogenism like severe hirsutism or severe acne
* Presence or a history of venous or arterial thrombotic/thromboembolic events (e.g., deep venous thrombosis, pulmonary embolism, myocardial infarction) or of a cerebrovascular accident.
* Presence or history of prodromi of a thrombosis (e.g., transient ischaemic attack, angina pectoris).
* History of migraine with focal neurological symptoms.
* Diabetes mellitus with vascular involvement.
* Presence of a severe or multiple risk factor(s) for venous or arterial thrombosis
* Pancreatitis or a history thereof if associated with severe hypertriglyceridemia
* Presence or history of severe hepatic disease as long as liver function values have not returned to normal.
* Presence or history of liver tumors (benign or malignant).
* Known or suspected sex-steroid influenced malignancies (e.g., of the genital organs or the breasts)
* Undiagnosed vaginal bleeding.
* Known or suspected pregnancy.
* Hypersensitivity to the active substances or to any of the excipients.
* Body-mass index (BMI ) more than 30.0 kg/m²
* Hypersensitivity to any of the study drug ingredients
* Any disease or condition that can compromise the function of the body systems and could result in altered absorption, excessive accumulation, impaired metabolism, or altered excretion of the study medication
* Known current or history of alcohol or drug abuse
* Prohibited concomitant medication:

  * Use of additional steroid hormones, anticoagulants (e.g., heparin, coumarin), antiepileptics (hydantoin derivates, e.g., phenytoin or carboxamide derivates, e.g., carbamazepin, oxcarbamazepin), other antiepileptics, (e.g., Felbamate, Topiramate), hypnotic and sedative (e.g., barbiturate derivates, primidone), tuberculostatics (e.g., rifampicin), oral antimycotics (e.g., griseofulvin, ketoconazole, itraconazole, fluconazol), virostatic agents (e.g., ritonavir), and products containing St. John's wort and continuous systemic use of antibiotics.
  * Medication with influence on libido (e.g., antihypertensives like beta-adrenergic blocker, cholinesterase blocking agents), psychotropic drugs (e.g., antidepressants, neuroleptic agents, selective serotonin reuptake inhibitors [SSRIs]), lipid lowering drugs and H2 blockers.
* Intake of an experimental drug within 3 months prior to inclusion in the study
* Previous assignment to treatment (e.g., randomization) during this study
* Close affiliation with the investigational site; e.g., a close relative of the investigator, dependent person (e.g., employee or student of the investigational site).
* Operation scheduled in the study period
* Abnormal laboratory values within the non-inclusion range
* Patient is in custody by order of an authority or a court of law

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2007-11; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
FSDS questionnaire (sexual desire and arousal component scores) | at baseline and after Cycle 6

SECONDARY OUTCOMES:
Change from baseline period to cycle 6 in the number of satisfactory sexual events | after Cycle 6
FSFI questionnaire (absolute values and change from baseline) - All domains | Cycle 1, 3, 6 and follow-up
FSDS-R questionnaire results | Cycle 1, 3, 6 and follow-up
FSEP questionnaire results | Cycle 1, 3, 6 and follow-up
PGWBI questionnaire results | Cycle 1, 3, 6 and follow-up
Serum hormone levels (SHBG, T, DHEA, DHEA-S) | Cycle 1, 3, 6 and follow-up
Vaginal pH | Cycle 1, 3, 6 and follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (2):
- Germany (2):
  - Hamburg, Hamburg
  - Berlin, State of Berlin

REFERENCES:
- See also: Click here and search for Bayer products information provided by the EMA — http://www.clinicaltrialsregister.eu